CLINICAL TRIAL: NCT03728049
Title: Point-of-care Haemostasis Testing of Von Willebrand Factor Function Embedded in Catheterization Laboratory to Improve Real-time Management of Paravalvular Regurgitation During Minimally Invasive TAVI
Brief Title: Von Willebrand Factor Point-of-care Testing to Improve Minimally Invasive TAVI Outcomes
Acronym: WITAVI-REAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Siemens Healthineers, France (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017_77; 2018-A01175-50 (Other: ID-RCB number, ANSM); PHRC-17-0697 (Other: PHRC number, DGOS)
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-05

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: Transcatheter Aortic Valve Replacement; Paravalvular regurgitation; Point-of-care test; Biomarker; Aortic stenosis; Von willebrand Factor
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Multicenter open-label randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-ADP group (Experimental): PVR assessment with the standard methods and with the CT-ADP that will be provided to the operator in real-time during TAVI. The decision to undertake corrective procedure will be left at the discretion of the operator and based on the results of the CT-ADP on top of the standard methods of PVR assessment.
  Interventions: Diagnostic Test: CT-ADP performed during TAVI procedure
- Control group (Other): PVR assessment with standard methods only (at discretion of the operator excluding CT-ADP and transesophageal echocardiography). CT-ADP will not be provided to the operator at the time of TAVI. The decision to undertake corrective procedure will be left at the discretion of the operator according to the results of the standard methods of PVR assessment.
  Interventions: Other: No CT-ADP performed during TAVI procedure

INTERVENTIONS:
Diagnostic Test: CT-ADP performed during TAVI procedure — The CT-ADP will be performed in the catheterization laboratory and revealed to the operator. The decision to undertake corrective procedure will be based on CT-ADP on top of standard methods of PVR assessment.
  Arms: CT-ADP group
Other: No CT-ADP performed during TAVI procedure — PVR assessment with the standard methods only (TTE and/or angiography and/or hemodynamics but excluding TEE and CT-ADP). The decision to undertake corrective procedure will be left at the discretion of the operator.
  Arms: Control group

SUMMARY:
Paravalvular regurgitation (PVR) is an important complication of Transcatheter Aortic Valve Implantation (TAVI) that is associated with a 2.5-fold increase risk of mortality. Transesophageal echocardiographic (TEE) is considered as the gold standard to assess the severity of PVR and guide the physician to perform corrective procedures during TAVI, but it requires general anesthesia (GA). With such approach (TEE+GA), the PARTNERII trial has demonstrated that very low rate of PVR (3,5%) can be achieved with current devices. Registries have demonstrated a strong trend for using a mini-invasive approach in which the procedure is performed under conscious sedation (CS) without TEE. However, several studies raised concerns on the safety of this mini-invasive approach concerning the PVR rate. Thus, the accurate and real-time assessment of the presence and severity of PVR is an unmet clinical need to optimize TAVI without TEE guidance. A recent study reported that a blood biomarker reflecting the Von Willebrand factor (VWF) activity, i.e. the closure time with adenosine diphosphate (CT-ADP), is a valuable non-invasive, highly reproducible, and easy to perform alternative to TEE for PVR evaluation.

The hypothesis is that the measurement of CT-ADP during TAVI performed without TEE guidance can improve both the detection of significant PVR and thus the procedural and clinical outcomes (primary objective).

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to undergo mini-invasive TAVI at any of the participating centers and fulfilling the inclusion criteria will be eligible for entry in the study. The decision to undertake TAVI will be made by the local heart team.
* Symptomatic aortic stenosis scheduled to undergo TAVI
* TAVI performed via mini-invasive approach defined as: transfemoral access route; local anesthesia/conscious sedation; no TEE guidance.
* All types of prosthetic valves (balloon-expandable, self-expandable, others) are accepted

Exclusion Criteria:

* TAVI through non-transfemoral approach
* TAVI with concomitant percutaneous coronary intervention
* TAVI performed under general anesthesia
* TAVI performed under TEE guidance
* Valve-in-valve procedure
* Inability to provide informed consent
* Associated ≥ moderate mitral regurgitation
* Peri-procedural treatment with ticagrelor or prasugrel treatment / direct oral anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 944 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
composite 1-year event rate of | At 1 year
  rate of All-cause death; rate of Paravalvular regurgitation ≥ moderate; rate of Rehospitalization; rate of Stroke; rate of Delayed valve re-intervention; rate of Mean transaortic gradient >20mmHg.

SECONDARY OUTCOMES:
All-cause death rate | At 30 days, at 1 year
  All-cause death
PVR rate | At 30 days, at 1 year
  PVR superior or egal to moderate
Rehospitalization for heart failure rate | At 30 days, at 1 year
  Rehospitalization for heart failure
Delayed valve re-intervention rate | At 1 year
  Delayed valve re-intervention
Delayed valve re-intervention rate | At 30 days, at 1 year
  Delayed valve re-intervention
Mean transaortic gradient >20mmHg rate | At 30 days
  Mean transaortic gradient >20mmHg
composite event rate | At 30 days
  All-cause death; PVR superior or egal to moderate; Rehospitalization for heart failure; All stroke (transient or definite); Delayed valve re-intervention; Mean transaortic gradient >20mmHg
composite event rate of the following individual safety endpoints | at 24hours
  Aortic injury; Coronary artery occlusion; Tamponade; All stroke (transient or definite)
Aortic injury rate | at 24hours
  Aortic injury
Coronary artery occlusion rate | at 24hours
  Coronary artery occlusion
Tamponade rate | at 24hours
  Tamponade
All stroke (transient or definite) rate | at 24hours
  All stroke (transient or definite)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vanbelle, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (9):
- France (9):
  - Hopital Estaing - Chu63 - Clermont Ferrand, Clermont-Ferrand
  - Institut Coeur-Poumon, CHU, Lille
  - Chu Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - Hu Pitie Salpetriere Aphp - Paris 13, Paris
  - Hopital Haut-Leveque - Chu - Pessac, Pessac
  - Chru Rennes Site Pontchaillou, Rennes
  - Hopital Civil / Nouvel Hopital Civil - Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse